CLINICAL TRIAL: NCT02958852
Title: A Clinical Trial to Compare Efficacy and Tolerability of Atorvastatin in Addition to Endocrine Treatment With Focus on Mechanisms of Resistance to Endocrine Treatment (Fulvestrant/Aromatase Inhibitors) in Patients With Advanced Breast Cancer
Acronym: ABC-SE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: South Sweden Breast Cancer Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OKFE 15-ABC-SE
Record Dates: First submitted 2016-10-05; First posted 2016-11-08 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Endocrine Treatment; Atorvastatin; Mechanisms of Resistance; Statins; Fulvestrant; Circulating Tumor Cells; Statins and Endocrine Treatment; Tumor Marker Expression; ER+ Metastatic Breast Cancer; Circulating Tumor DNA; Cholesterol
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Letrozole; Atorvastatin; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Letrozole (Active Comparator): Confirmed ER positive/HER2 negative metastatic breast cancer, including locally advanced stage IV disease, requiring systemic endocrine treatment, in this case letrozole, 2.5 mg daily until progression of disease. Upon progression of first line, patients will receive second line treatment using fulvestrant.
  Interventions: Drug: Letrozole
- Letrozole+Atorvastatin (Experimental): Confirmed ER positive/HER2 negative metastatic breast cancer, including locally advanced stage IV disease, requiring systemic endocrine treatment, in this case letrozole, 2.5 mg daily, with the addition of atorvastatin, 40 mg daily until progression of disease. Upon progression of first line, patients will receive second line treatment using fulvestrant.
  Interventions: Drug: Letrozole and atorvastatin
- Fulvestrant (Other): Fulvestrant will be used as second line endocrine treatment upon progression on first line with letrozole +/- atorvastatin.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Letrozole — Daily orally
  Arms: Letrozole
Drug: Letrozole and atorvastatin — Daily orally
  Arms: Letrozole+Atorvastatin
Drug: Fulvestrant — Fulvestrant will be used as second line treatment upon progression on first line treatment with letrozole +/- atorvastatin.
  Arms: Fulvestrant

SUMMARY:
A Clinical Trial to Compare Efficacy and Tolerability of Atorvastatin in Addition to Endocrine Treatment with Focus on Mechanisms of Resistance to Endocrine Treatment (fulvestrant/aromatase inhibitors) in Patients With Advanced Breast Cancer.

DETAILED DESCRIPTION:
A randomized, open-labelled, phase II trial in the first and second-line metastatic treatment setting, comparing standard endocrine treatment (aromatase inhibitor (AI)) with endocrine treatment plus atorvastatin (1:1). Upon progression in the first line setting, and as part of the translational studies on mechanisms of resistance to endocrine therapy, the patients will receive second line endocrine treatment using fulvestrant. Upon progression to first line treatment, patients that were receiving atorvastatin will stop this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women with confirmed ER positive/HER2 negative metastatic breast cancer, including locally advanced stage IV disease, requiring systemic endocrine treatment.
2. Age > 18 years.
3. Performance status of Eastern Cooperative Oncology Group (ECOG) ≤ 2.
4. Metastatic disease must be radiologically or clinically assessable, by means of at least one of the following techniques: clinical examination, computerized tomography (CT), magnetic resonance imaging (MRI), bone scintigraphy or positron emission tomography (PET). Bone metastases alone are allowed.
5. Pre-menopausal patients must consent to undergo either surgical or chemical castration during the duration of the treatment and utilize an effective contraception barrier method.
6. Patient not willing to undergo study specific biopsy from the metastatic site should preferably have enough metastatic tumor sample material archived to perform RNA extraction from formalin fixed paraffin embedded (FFPE) material.
7. Patient must be capable and willing to grant signed informed consent prior to any procedure related with this study as well as to allow access to FFPE biopsies for RNA extraction and for serial circulating tumor cells capture. Biopsy of the metastatic site upon progression is not mandatory but desirable.
8. Signed informed consent according to International Conference on Harmonization /Good Clinical Practice, and national/local regulations.
9. Patients currently on first-line treatment with an AI for metastatic breast cancer who cannot participate on the first part of the treatment (taking lowering cholesterol drugs, or already on AIs for metastatic disease when study is opened) can be eligible to enter on the second part to study mechanisms of resistance to fulvestrant once they have progressed to AI.
10. Patients that progress while taking AI as adjuvant treatment, have confirmed hormone receptor+ metastatic breast cancer and are not deemed suitable for first line AI will also be eligible to enter directly in the second part of the study and be treated with fulvestrant up-front.

Exclusion Criteria:

1. Previous treatment for metastatic breast cancer (previous systemic treatment for early breast cancer allowed), unless being considered for direct entry to the second part of the study with fulvestrant (see inclusion criteria 9 and 10).
2. Brain as the only site of metastatic breast cancer.
3. Ongoing treatment with statins (e.g. simvastatin, atorvastatin, fluvastatin, lovastatin, pravastatin, or rosuvastatin), anion-exchangers (e.g. colestyramin or colesevelam), fibrates (e.g. gemfibrozil), nicotin-acids (or acipimox) or inhibitors of intestinal cholesterol uptake (e.g.ezetimibe ) for the first part of the trial.
4. Evidence of hepatic dysfunction (alanine aminotransferase level more than three times the upper limit of the normal range) or renal dysfunction (creatine kinase level) more than three times the upper limit of the normal range.
5. Known coagulation disorders or treatment with a 4-hydroxycoumarin derivative is an exclusion criterion for the fulvestrant treated patients.
6. Treatment with anticoagulants other than 4-hydroxycoumarin derivatives or antiplatelet drugs. Patients in treatment with heparin can interrupt treatment 24h prior to biopsies and resume treatment 12h after biopsy has been performed. In case of patients treated with clopidogrel or salicylates, they should be able to interrupt treatment 5-7 days before biopsy and resume 24h after.
7. History of hemorrhagic stroke.
8. Pregnancy or breast-feeding.
9. Untreated psychiatric disorders that will impair the patient's ability to comply with study treatment or protocol.
10. History of allergic reactions attributed to compounds of similar chemical or biological composition to either of the study drugs.

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate. | 6 months after the last patient has been randomly assigned.
  Clinical benefit rate (CBR), defined as the proportion of all randomly assigned patients who have the best overall response a complete response, a partial response, or stable disease up to 24 weeks following first-line letrozole treatment alone or in combination with atorvastatin.

SECONDARY OUTCOMES:
Progression free survival. | 6 months after the last patient has been randomly assigned. Data cut off, 15th October 2020.
  Progression free survival (PFS) comparing endocrine treatment alone or endocrine treatment in combination with atorvastatin in patients with advanced breast cancer. It is defined as the time elapsing between the time of random assignment to treatment and the date of the earliest evidence of objective disease progression or death of any cause before documented disease-progression assessed through study completion.
Objective response rate. | 6 months after the last patient has been randomly assigned. Data cut off, 15th October 2020.
  Objective Response Rate (ORR; the proportion of patients with a best overall response of either a complete response or a partial response) through study completion.
Time to progression. | From date of treatment start until the date of first documented progression. Data cut off, 15th October 2020.
  Time-To-Progression (TTP) defined as time elapsed between date of diagnosis of metastatic disease and date of confirmation of disease progression in the first part of the protocol assessed through study completion. The primary analysis will be performed 6 months after the last patient has been randomly assigned.
Duration of Clinical benefit. | 6 months after the last patient has been randomly assigned. Data cut off, 15th October 2020.
  Duration of Clinical Benefit (DCB) includes complete response, partial response and disease stabilization assessed through study completion.
Overall survival. | 6 months after the last patient has been randomly assigned. Data cut off, 15th October 2020.
  Overall survival defined as the time elapsed from the date of first confirmation of metastatic disease and the date of death from any cause through study completion.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | From date of treatment start, until 1 month after the last patient in the study has finished the trial.
  Information regarding the number of participants with abnormal laboratory values and/or adverse events that are related to treatment is collected continuously during the trial assessed through study completion.
  Differences between treatment arms in incidence of recorded cardiovascular events and/or incident diabetes mellitus during and after study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Signe Borgquist, MD, PhD, Principal Investigator — Lund University Hospital, Department of Oncology
Locations (1):
- Lund University Hospital, Department of Oncology, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No